CLINICAL TRIAL: NCT02625415
Title: A Double Blind Placebo Control Randomised Trial to Test the Effectiveness of Vitamin B6 in Hand Foot Syndrome
Brief Title: The Topical Application of Vitamin B6 in Palmar-Plantar Erythrodysesthesia
Acronym: HFSB6
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyprus University of Technology (Other)
Collaborators: American Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Andreas Charalambous, Assistant Professor, Cyprus University of Technology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: AC-PPEHP-89
Record Dates: First submitted 2015-12-05; First posted 2015-12-09 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Palmar-Plantar Erythrodysesthesia
MeSH Terms: conditions — Hand-Foot Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin B6 (Experimental): Topical application of B6 cream to the hand or/and feet 1-2 ml applied to the hand or /and feet three times a day for 4 weeks.
  Interventions: Device: Vitamin B6 cream
- Placebo (Placebo Comparator): Topical application of B6 Placebo cream to the hand or/and feet 1-2 ml applied to the hand or /and feet three times a day for 4 weeks.
  Interventions: Device: Placebo Vitamin B6 cream

INTERVENTIONS:
Device: Vitamin B6 cream — Topical Vitamin B6 cream
  Arms: Vitamin B6
Device: Placebo Vitamin B6 cream — Placebo Vitamin B6 cream
  Arms: Placebo

SUMMARY:
The study is designed to test the effectiveness of topical B6 cream in patients that developed Palmar-Plantar Erythrodysesthesia (Hand foot syndrome).

DETAILED DESCRIPTION:
This will be a randomized double-blind, placebo-controlled study with 100 cancer patients that will receive chemotherapy treatment with capecitabine and/or pegylated liposomal doxorubicin. The selection of potential participants will be based on inclusion and exclusion criteria. Patients will be randomly allocated either to the treatment group or the placebo group. Treatment will be delivered daily (t.d.s) and assessments will take place at 0, 1, 2, 3 and 4 weeks.

The intervention group will receive the application of topical vitamin B6 cream to the hands and/or feet of the patients and the control group will receive the placebo.

At both baseline and follow-up, patients in both groups will be assessed for their degree of palmar-plantar erythrodysesthesia, the Quality of Life, the need for dose-limiting due to PPE and Pain intensity using standardized rating scales. Data will be analysed with inferential and descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

* Adult cancer patients (>18)
* Patients receiving capecitabine and/or PLD as monotherapy or in combination with other agents
* Patients that will experience PPE grade 1 or above
* Willing to participate
* Ability to complete the psychometric assessments.
* A performance status of two or less on the Eastern Cooperative Oncology Group (ECOG

Exclusion Criteria:

* Patients with hypersensitivity to Vitamin B.
* Patients with pre-existing dermatological condition affecting the hands or/and feet that may limit the interpretation of results
* Patients on oral Pyridoxine or nicotine patches
* Patients with a previous history of PPE
* Patients whose chemotherapy was discontinued for more than a week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-07; Primary Completion 2018-05-01 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
PPE grade | up to 4 weeks
  The grade of PPE will be assessed with a standardised three-grade system previously used in capecitabine clinical trials (Scheithauer et al 2003)

SECONDARY OUTCOMES:
Health Related Quality of Life | up to 4 weeks
  The HRQoL of the patients will be assessed with the EORTC QLQ -C30 module which has been developed and validated explicitly for patients suffering from cancer.
Quality of Life in relation to PPE | up to 4 weeks
  This is a quality of life scale specifically for patients experiencing radiation-induced PPE

OTHER OUTCOMES:
Activities of daily living | up to 4 weeks
  Activities of daily living will be assessed with the Eastern Co-operative Oncology Group (ECOG)/WHO system
Treatment side-effects | up to 4 weeks
  Any possible side-effect due to the treatment will be recorded

CONTACTS AND LOCATIONS:
Locations (2):
- Cyprus (2):
  - Limassol General Hospital, Limassol
  - American Medical Center, Nicosia

REFERENCES:
- [Derived] Charalambous A, Tsitsi T, Astras G, Paikousis L, Filippou E. A pilot randomized double-blind, placebo-controlled study on the effects of the topical application of pyridoxine on palmar-plantar erythrodysesthesia (PPE) induced by capecitabine or pegylated liposomal doxorubicin (PLD). Eur J Oncol Nurs. 2021 Feb;50:101866. doi: 10.1016/j.ejon.2020.101866. Epub 2020 Nov 11. PMID 33227569